CLINICAL TRIAL: NCT05854199
Title: THIS-WIC Telehealth Solutions: Evaluation With North Carolina WIC Clients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency); North Carolina Department of Health and Human Services (Other Government); RTI International (Other)
Responsible Party: Principal Investigator, Erin Hennessy, Assistant Professor, Division of Nutrition Interventions, Communication and Behavior Change Director ad interim, ChildObesity180 Friedman School of Nutrition Science and Policy, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00002935
Record Dates: First submitted 2023-05-02; First posted 2023-05-11 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Telehealth; Nutrition Education; Dietary Intake; WIC
Keywords: Telehealth; WIC; nutrition education; dietary intake

STUDY DESIGN:
Intervention Model Description: Study participants will be clients at local WIC agency sites where either the telehealth solution is offered or where only usual care is available (control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth solution (Experimental): Telehealth solution offered
  Interventions: Behavioral: Telehealth solution
- Usual care (No Intervention): Control

INTERVENTIONS:
Behavioral: Telehealth solution — Telehealth nutrition education platform
  Arms: Telehealth solution

SUMMARY:
With funding through the United States Department of Agriculture (USDA) and Tufts University's Telehealth Intervention Strategies for WIC (THIS-WIC) project, North Carolina (NC) WIC department will be implementing new, nutrition education telehealth in NC's WIC program. The purpose of this study is to evaluate the impact of the telehealth platform. The evaluation will focus on NC WIC clients as the study population. The North Carolina WIC department would be implementing this education platform, regardless of the evaluation research. The North Carolina WIC department is responsible for implementing this new intervention, while the Tufts University research team is responsible for the evaluation of this platform through surveys and analysis of administrative data.

An online survey will be used to gauge WIC clients' satisfaction with the telehealth solution and the impact of the telehealth solution compared to usual care on breastfeed duration, dietary intake, attendance at scheduled appointments, attitudes to breastfeeding and nutrition education, and barriers encountered. Survey data will be combined with previously collected data on clients and their families from the NC Management Information Systems (MIS), and aggregate level data from the telehealth solution about utilization.

DETAILED DESCRIPTION:
Telehealth can reduce barriers and increase access to care, and it can be applied to the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). WIC is a federal nutrition assistance program that helps low-income women with children up to age 5. There is a large volume of research that supports remote patient monitoring, and the most benefits are found when telehealth is used for communication and counseling. The USDA awarded Tufts University a grant to test and evaluate the use of telehealth innovations in the delivery of USDA's WIC program. Tufts University then offered the USDA/Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) grant opportunity to WIC state agencies across the US. THIS-WIC selected 7 WIC State Agencies to receive grants, and the NC state agency is one recipient. The THIS-WIC team at Tufts University is leading the evaluation of these telehealth solutions in collaboration with funded WIC State Agencies.

THIS-WIC aims to generate evidence from NC's telehealth solution to inform how the telehealth solution supports WIC services compared to usual in-person care. The NC telehealth platform includes a mobile-optimized website, meaning that it functions as an app without requiring the amount of memory and data that apps use. Evaluation findings will inform stakeholders about the platform's benefits and how viable it is to sustain and adapt more widely.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* postpartum women
* parent/guardian of a participating infant or child in the WIC program

Study participants will be clients at local WIC agency sites where either the telehealth solution is offered or where only usual care is available (control).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 892 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Satisfaction with the telehealth solution | During the study period, approximately 12 months
  WIC clients satisfaction with nutrition education offered via the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

SECONDARY OUTCOMES:
Breastfeeding duration | During the study period, approximately 12 months
  Duration of breastfeeding in clients offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attendance at scheduled appointments | During the study period, approximately 12 months
  WIC clients attendance at appointments when offered the telehealth solution compared to usual care. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Dietary intake | During the study period, approximately 12 months
  Impact of the telehealth solution compared to usual care on dietary intake. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Attitudes to breastfeeding and nutrition education | During the study period, approximately 12 months
  Impact of the telehealth solution compared to usual care on WIC clients' attitudes to breastfeeding and nutrition education. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.
Barriers encountered in obtaining nutrition education | During the study period, approximately 12 months
  Impact of the telehealth solution compared to usual care on barriers encountered by WIC clients in obtaining nutrition education. Data will be collected, and this outcome measure will be assessed via survey completion by study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Hennessy, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Tufts Telehealth Intervention Strategies for WIC (THIS-WIC) website — https://thiswic.nutrition.tufts.edu/